CLINICAL TRIAL: NCT03181997
Title: TOP-AS Registry: Transcatheter Aortic Valve Implantation in Oncology Patients With Severe Aortic Stenosis
Brief Title: Outcomes of Transcatheter Aortic Valve Implantation in Oncology Patients With Severe Aortic Stenosis
Acronym: TOP-AS
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Uri Landes, Principal Investigator, Rabin Medical Center
Other Study IDs: 0136-17-RMC
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Aortic Valve Stenosis; Malignancy
Keywords: Aortic Valve Stenosis; Transcatheter Aortic Valve Implantation; Cancer; Malignancy
MeSH Terms: conditions — Aortic Valve Stenosis; Neoplasms | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- TAVI Patients with active cancer: Patients with active cancer undergoing transcatheter aortic valve implantation (TAVI) with native aortic valves.
  Interventions: Device: Native aortic valve; Procedure: Transcatheter aortic valve implantation (TAVI)
- TAVI patients without cancer: Patients with no active cancer undergoing transcatheter aortic valve implantation (TAVI) with native aortic valves.
  Interventions: Device: Native aortic valve; Procedure: Transcatheter aortic valve implantation (TAVI)

INTERVENTIONS:
Device: Native aortic valve — Native valve, with any transcatheter heart valve type
Procedure: Transcatheter aortic valve implantation (TAVI) — Percutaneous aortic valve implantation preformed in one of these methods: transfemoral, transapical,subclavian or other.

SUMMARY:
As for today, transcatheter aortic valve implantation (TAVI) is indicated only in symptomatic patients with severe aortic stenosis (AS) at high surgical risk. As cancer therapy improves, some AS patients suffering active malignancy (including advanced metastatic diseases) may be more endangered by their untreated valvular disease than their oncological disease. Among these patients, TAVI may be indicated before cancer related surgery or cardiotoxic anti-cancer therapy in order to achieve better anti-cancer therapy outcomes. Individualized life expectancy assumptions should be evaluated by the heart team in the clinical decision-making process as an essential factor in weighing the risk-benefit ratio for oncologic patients undergoing TAVI. A multicenter, international TAVI in Oncology Patients with AS (TOP-AS) registry was designed to collect data on patients with an active malignancy and severe AS undergoing TAVI. The aim of the study is to evaluate the outcomes, benefits and risks of oncology patients undergoing TAVI, mainly the patients' survival and cause of death and also the interactions between the valvular and the oncologic conditions.

DETAILED DESCRIPTION:
The TAVI program was initiated in Rabin Medical Center in 2008 and the institutional review board approved the prospective collection of our TAVI Database (i.e. RECORD TAVI). During these years, several oncology patients were treated with TAVI. Also, in daily practice a few asymptomatic AS patients in whom TAVI was indicated before cancer related surgery / cardiotoxic anti-cancer therapy underwent TAVI.

This study will initiate a multicenter, international registry designed to collect data on TAVI in cancer patients in correspondence to medical records within each center. Data will be collected retrospectively for cases performed before registry initiation and prospectively thereafter. All inconsistencies regarding data collection will be resolved directly with local investigators and on-site data monitoring. Patients' inclusion approval is by a local ethics committee in each center.

Saving Data: Data will be recorded in Excel table; each center and patient will receive a unique code so the data file will be anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active malignancy (all types excluding non-melanoma skin Ca)
* Severe aortic stenosis undergoing native valve TAVI (any transcatheter heart valve type).

Exclusion Criteria:

* TAVI for conditions other than severe AS.
* Valve in valve TAVI patient.
* Patients cured /in remission from cancer during the index TAVI.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be selected from several international transcatheter aortic valve implantation centers.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Patients survival | 2 years
  Patients survival in days

SECONDARY OUTCOMES:
New York Heart Association Functional Classification (NYHA FC) | 2 years
  Provides information regarding patients functional status on scale of 1-4.
Cause of death | 2 years
  Whether the cause of death is cardiovascular or non-cardiovascular.

CONTACTS AND LOCATIONS:
Overall Officials: Ran Kornowski, Prof,MD, Study Chair — Chairman, Dept. of Cardiology, Rabin Medical Center, Israel; Ran Kornowski, Prof,MD, Study Director — Chairman, Dept. of Cardiology, Rabin Medical Center, Israel; Uri Landes, MD, Principal Investigator — Dept. of Cardiology, Rabin Medical Center, Israel
Locations (1):
- Rabin Medical Center,, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swain SM, Kim SB, Cortes J, Ro J, Semiglazov V, Campone M, Ciruelos E, Ferrero JM, Schneeweiss A, Knott A, Clark E, Ross G, Benyunes MC, Baselga J. Pertuzumab, trastuzumab, and docetaxel for HER2-positive metastatic breast cancer (CLEOPATRA study): overall survival results from a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Oncol. 2013 May;14(6):461-71. doi: 10.1016/S1470-2045(13)70130-X. Epub 2013 Apr 18. PMID 23602601
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Fleisher LA, Jneid H, Mack MJ, McLeod CJ, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A. 2017 AHA/ACC Focused Update of the 2014 AHA/ACC Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2017 Jul 11;70(2):252-289. doi: 10.1016/j.jacc.2017.03.011. Epub 2017 Mar 15. No abstract available. PMID 28315732
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Guyton RA, O'Gara PT, Ruiz CE, Skubas NJ, Sorajja P, Sundt TM 3rd, Thomas JD; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC guideline for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jun 10;63(22):e57-185. doi: 10.1016/j.jacc.2014.02.536. Epub 2014 Mar 3. No abstract available. PMID 24603191
- [Derived] Landes U, Iakobishvili Z, Vronsky D, Zusman O, Barsheshet A, Jaffe R, Jubran A, Yoon SH, Makkar RR, Taramasso M, Russo M, Maisano F, Sinning JM, Shamekhi J, Biasco L, Pedrazzini G, Moccetti M, Latib A, Pagnesi M, Colombo A, Tamburino C, D' Arrigo P, Windecker S, Pilgrim T, Tchetche D, De Biase C, Guerrero M, Iftikhar O, Bosmans J, Bedzra E, Dvir D, Mylotte D, Sievert H, Watanabe Y, Sondergaard L, Dagnegard H, Codner P, Kodali S, Leon M, Kornowski R. Transcatheter Aortic Valve Replacement in Oncology Patients With Severe Aortic Stenosis. JACC Cardiovasc Interv. 2019 Jan 14;12(1):78-86. doi: 10.1016/j.jcin.2018.10.026. PMID 30621982